CLINICAL TRIAL: NCT03647033
Title: Phacoemulsification Versus Phacoemulsification With Micro-bypass Stent Implantation in Primary Angle Closure and Primary Angle Closure Glaucoma: Randomized Double-masked Clinical Trial
Brief Title: Phacoemulsification Versus Phacoemulsification With Micro-bypass Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khoo Teck Puat Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/00644
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-09

CONDITIONS: Primary Angle-Closure Glaucoma; Primary Angle Closure Without Glaucoma Damage
Keywords: istent; primary angle closure
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Intervention Model Description: Single centre, randomised prospective trial, the patient and the intraocular pressure (IOP)checking staff will be blinded. Randomised by random envelope shuffle technique.
  1:1 ratio allocation 2 arms: phacoemulsification alone and phacoemulsification and iStent. 16 patients in each arm, 32 patients in total. The post-operative management is the same for both arms After operation the patient will be followed up at day 1, week 1, week 2, months 1, 3, 6 and 12.
  At each visit the patient will have the following tests: Tonometry (IOP check) - Not to be taken by the operating surgeon, to be taken by 2 people, one IOP checker and one reader.
Who Masked: Participant, Outcomes Assessor
Masking Description: Shuffled envelope system. Patient will be blinded to the procedure. The intraocular pressure (IOP) measure and reader will be blinded to the procedure.
  There will be no planned breaking of randomization. Unplanned breaking will happen if any envelopes are damaged or lost. Unmasking will take place after 1 year post operation by the study team to inform the patient of the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- phacoemulsification alone (No Intervention): routine phacoemulsification cataract surgery with intraocular lens implantation
- phacoemulsification and iStent (Experimental): phacoemulsification cataract surgery with intraocular lens implantation combined with iStent implantation
  Interventions: Device: iStent implantation

INTERVENTIONS:
Device: iStent implantation — The iStent is a FDA and Health Sciences Authority (HSA) approved micro-bypass stent device that bypasses the trabecular meshwork (filtration membrane of the aqueous fluid exit pathway) and reroutes aqueous from the anterior chamber directly into canal of Schlemm and out of the eye. It lowers the intraocular pressure (IOP) by increasing the outflow of fluid from the eye from the micro-bypass. In angle closure, the lens has to be removed to create enough space for the iStent to be inserted.
  Arms: phacoemulsification and iStent

SUMMARY:
Assessing the safety and efficacy of a micro-bypass stent in combination with cataract surgery in subjects with primary angle closure. Subjects are randomized into two arms: phacoemulsification cataract surgery alone versus phacoemulsification cataract surgery combined with the micro-bypass stent implantation. Post surgery intraocular eye pressure will be recorded to assess the efficacy of both arms.

DETAILED DESCRIPTION:
Aim: To assess the safety and efficacy of the iStent trabecular micro-bypass stent (Glaukos Corporation, Laguna Hills, CA) in combination with cataract surgery in subjects with primary angle closure and mild to moderate primary angle closure glaucoma

Method: Prospective, randomised controlled trial, blinded to patient and intra-ocular pressure measuring staff. 32 patients, 1:1 ratio, in 2 arms of phacoemulsification alone compared to phacoemulsification with iStent.

Hypothesis: Phacoemulsification with micro-bypass stent has a better intraocular pressure (IOP) lowering effect compared to phacoemulsification alone in primary angle closure and primary angle closure glaucoma at 1 year after surgery.

Importance: Primary angle closure and primary angle closure glaucoma are conventionally treated with eye drops that lower the intraocular pressure (IOP). Phacoemulsification/lens extraction can often help lower the eye pressure by widening the drainage angle and via ultrasound mechanisms, however, in some cases the IOP is not lowered, or even can cause the IOP to be higher. The iStent implant can be used together with phacoemulsification to lower the IOP and in Primary open angle glaucoma, it gives an additional 20% IOP reduction. It is unclear what effect the iStent has in primary angle closure or primary angle closure glaucoma as it has never been studied. It is important because primary angle closure glaucoma is much more common in the Singaporean Chinese population and the iStent can potentially be used to control the IOP instead of conventional eye drops and glaucoma surgery which have their own potential adverse effects.

Potential Benefits: iStent with phacoemulsification may control the IOP better than phacoemulsification alone, reduce the need for IOP lowering medication after surgery, and prevent the need for glaucoma surgery in the future.

Potential Risks: The iStent has risks of IOP spikes, bleeding in the anterior chamber and iStent dislocation.Phacoemulsification has the risks of: infection, bleeding, reduced vision, inflammation, posterior capsular rupture, vitreous loss, retinal detachment, endophthalmitis, suprachoroidal haemorrhage and Intraocular Lens dislocation.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* Previous diagnosis of Primary Angle Closure or Primary Angle Closure Glaucoma
* Intraocular Pressure above 21mmHg at 3 separate visits
* On 1 or more hypotensive medications
* Pre-operative visual acuity of no better than 6/12

Exclusion Criteria:

* Other glaucoma diagnosis: Primary Open Angle Glaucoma, secondary glaucoma
* Peripheral Anterior Synechiae in the nasal and inferior quadrant
* Cloudy cornea affecting view for iStent implantation
* Previous glaucoma surgery
* History of Ocular trauma
* Ocular surface disease
* Pre-proliferative or proliferative diabetic retinopathy
* Age related macular degeneration with macular scar or macular atrophy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2017-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philemon Huang, MMed, FAMS, Principal Investigator — National Healthcare Group, Singapore
Locations (1):
- Khoo Teck Puat Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Craven ER, Katz LJ, Wells JM, Giamporcaro JE; iStent Study Group. Cataract surgery with trabecular micro-bypass stent implantation in patients with mild-to-moderate open-angle glaucoma and cataract: two-year follow-up. J Cataract Refract Surg. 2012 Aug;38(8):1339-45. doi: 10.1016/j.jcrs.2012.03.025. PMID 22814041
- [Background] Fea AM. Phacoemulsification versus phacoemulsification with micro-bypass stent implantation in primary open-angle glaucoma: randomized double-masked clinical trial. J Cataract Refract Surg. 2010 Mar;36(3):407-12. doi: 10.1016/j.jcrs.2009.10.031. PMID 20202537
- [Background] Malvankar-Mehta MS, Iordanous Y, Chen YN, Wang WW, Patel SS, Costella J, Hutnik CM. iStent with Phacoemulsification versus Phacoemulsification Alone for Patients with Glaucoma and Cataract: A Meta-Analysis. PLoS One. 2015 Jul 6;10(7):e0131770. doi: 10.1371/journal.pone.0131770. eCollection 2015. PMID 26147908
- [Background] Samuelson TW, Katz LJ, Wells JM, Duh YJ, Giamporcaro JE; US iStent Study Group. Randomized evaluation of the trabecular micro-bypass stent with phacoemulsification in patients with glaucoma and cataract. Ophthalmology. 2011 Mar;118(3):459-67. doi: 10.1016/j.ophtha.2010.07.007. Epub 2010 Sep 15. PMID 20828829

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phacoemulsification Alone | Phacoemulsification and iStent
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phacoemulsification Alone | Phacoemulsification and iStent | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [64.3 to 76.8] | 65 [62 to 67] | 67 [63 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 7 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 16 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure Between Baseline and 1 Year
Description: change in mean unmedicated intraocular pressure between baseline and 1 year
Time Frame: 1 year
Population: intraocular pressure of participants measured in mmHg
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phacoemulsification Alone | Phacoemulsification and iStent
Number analyzed (Participants) | 16 | 16
mmHg | 15 (2.5) | 14.7 (3.1)

2. Secondary Outcome: Change in Glaucoma Medications
Description: change in number of topical glaucoma medications at 1 year post operation
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: number of glaucoma medications
Arm/Group | Phacoemulsification Alone | Phacoemulsification and iStent
Number analyzed (Participants) | 16 | 16
number of glaucoma medications | 0.75 (1.0) | 0.25 (0.68)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Phacoemulsification Alone | Phacoemulsification and iStent
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 10/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phacoemulsification Alone (N=16) | Phacoemulsification and iStent (N=16)
intraoperative hyphema (Eye disorders) | 0 (0) | 6 (6)
intraoperative iris prolapse (Eye disorders) | 1 (1) | 2 (2)
intraoperative iris trauma (Eye disorders) | 1 (1) | 1 (1)
intraoperative iridodialysis (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-10-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03647033/Prot_002.pdf
  • Informed Consent Form (2015-10-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03647033/ICF_003.pdf